CLINICAL TRIAL: NCT04884854
Title: Early Efferon LPS Hemoperfusion Through Hypercrosslinked Styrene-divinylbenzene Copolymer With Immobilized LPS-selective Ligand for Treatment of Patients With Septic Shock
Brief Title: Efferon LPS Hemoperfusion for Treatment of Patients With Septic Shock
Status: Completed | Type: Observational
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Other Study IDs: efferon-lps-2020-01
Record Dates: First submitted 2021-04-26; First posted 2021-05-13 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Septic Shock
Keywords: septic shock; extracorporeal therapy; LPS sequestration; abdominal sepsis
MeSH Terms: conditions — Shock, Septic; Intraabdominal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Efferon LPS — Efferon LPS is a single-use therapeutic device for extracorporeal blood purification using direct hemoperfusion. Detoxification is carried out by selective adsorption of lipopolysaccharides (bacterial endotoxins) and non-selective removal of cytokines by internal porous structure. It is a cylindrical polycarbonate casing filled with spherical granules of LPS-selective polymeric adsorbent mesoporous beads and isotonic sodium chloride solution. The device is registered in Russia as a medical device RZN 2019/8886.

SUMMARY:
Sepsis is a global healthcare burden sepsis, it reaches 20-30 million cases annually (WHO data). Numerous studies have shown that extracorporeal hemoperfusion therapies that eliminate endotoxin and\or excess of cytokines improve treatment outcomes in patients with septic shock. Aim of the study: to evaluate safety and feasibility of clinical use of an extracorporeal blood adsorber based on a hypercrosslinked styrene-divinylbenzene copolymer with immobilized lipopolysaccharide (LPS)-selective ligand designed to remove endotoxins from the bloodstream to treat patients with septic shock.

DETAILED DESCRIPTION:
Introduction. Sepsis, according to the latest consensus deﬁnition (SEPSIS-3, 2016), is a disease characterized by life-threatening organ failure resulting from a disordered regulation of the body's response to infection. Sepsis continues to be the leading cause of death in intensive care units in almost any country in the world.

The highest mortality rate in sepsis is associated with the development of septic shock (SS). Septic shock is deﬁned as sepsis (according to the criteria of SEPSIS-3, 2016) accompanied by severe hemodynamic, cellular and metabolic disorders, with a higher risk of fatal outcome than sepsis without shock. On average, SS is detected with a frequency of 8.3-10.4% among ICU patients, and its mortality, according to recent estimates, reaches 38-50% and even higher, exceeding 50-80% with such comorbidity as diabetes mellitus.

Success in treating septic shock is traditionally associated with adequate vasopressor, antibacterial, and anti-shock therapy, including inotropic support. At the same time, such factors as multiple antibiotic resistance of Gram-negative bacteria, changes in the intestinal microbiota and associated proﬁle of bacterial metabolites entering circulation and participating in the pathogenesis of sepsis, other bacterial products such as pathogen-associated molecular patterns and cytokines induced by them, bacterial endotoxins contributing most to the multiorgan failure, nowadays are considered as new targets for developing eﬀective mtools of controlling the septic shock sequelae.

Taking into account the key role of bacterial endotoxins in the pathogenesis of septic shock and the absence of a signiﬁcant trend for reducing mortality in response to the medication treatment, increasing interest is being focused on extracorporeal methods of clearing the endotoxins and inﬂammatory immune mediators from the bloodstream. Such methods are designed to reduce the levels of pathogenetically signiﬁcant molecules in the systemic circulation down to less critical values at least for a certain period of time in order to enable the immune system and antibiotics to reduce the bacterial load and the production of new endotoxin molecules.

The methods used and developed with respect to selective adsorption of endotoxin molecules from the bloodstream are promising. They provide, at early stages of the disease, interruption of the pro-inﬂammatory cascade initiated by inborn immune cells and causing organ dysfunction. At the same time, the place of LPS-selective hemoperfusion in sepsis therapy is still not clearly deﬁned.

Recently, the ﬁrst clinical experience of using a new generation of Eﬀeron LPS medical device for successful treatment of a patient with sepsis has been reported [Ushakova N.D., Tikhonova S.N., Rozenko D.A. Hemosorption by a Column Adsorber Based on Hyper-Cross-Linked Styrene-Divinylbenzene Copolymer with Immobilized Lipopolysaccharide-Selective Ligand in Combined Intensive Care of Lung Cancer-Related Postoperative Acute Lung Injury (Case Report). Obshchaya Reanimatologiya=General Reanimatology. 2020; 16 (4): 14-20. [In Russ.] DOI: 10.15360/1813-9779-2020-4-14-20].

This extracorporeal adsorber contains a multimodal sorbent based on a hypercrosslinked styrene-divinylbenzene copolymer with a covalently immobilized ligand to the Lipid A domain of LPS molecule. The combination of a porous matrix containing mesopores and ligand provides selective and simultaneous action of the adsorbent on two types of dissimilar therapeutic targets (cytokines and endotoxins, respectively).

Efferon LPS (Efferon JSC, Moscow, Russia) is a single-use therapeutic device for extracorporeal blood purification using direct hemoperfusion. Detoxification is carried out by selective adsorption of lipopolysaccharides (bacterial endotoxins) and non-selective removal of cytokines by internal porous structure. It is a cylindrical polycarbonate casing filled with spherical granules of LPS-selective polymeric adsorbent mesoporous beads and isotonic sodium chloride solution. The device is registered in Russia as a medical device RZN 2019/8886.

The aim of the study was to evaluate the safety and clinical eligibility of a novel medical device based on a hypercrosslinked styrene divinylbenzene copolymer with an immobilized LPS-selective ligand designed to remove endotoxins from the bloodstream for treatment of patients with septic shock.

Materials and methods. Nine patients (mean age 58 years, 5 men and 4 women, initial median APACHE II score 28 points, SOFA score 10 points) with confirmed gram-negative bacterial infection and septic shock (SEPSIS-3, 2016) underwent LPS-selective hemoperfusion using Efferon LPS for 6 hours, followed by prolonged venous-venous hemodiafiltration. The decision to use LPS-selective hemoperfusion in a particular patient was made by the attending doctor with the participation of a medical consultant team in accordance with clinical indications.

Before hemoperfusion (day 0), immediately after it, one day after its end (day 1) and once a day for the next 4 days, patients were determined hemodynamic parameters, oxygenation, signs of organ failure, leukocyte count, procalcitonin levels, C- reactive protein, IL 1β, clinical chemistry parameters. All patients underwent a test for endotoxin activity at the same time. Endotoxin Activity Assay Kit (EAA TM) (Spectral Medical Inc., Canada; Certiﬁcate No. FSZ 2009/04982) was used to determine endotoxin activity (EAA) using chemiluminescent rapid test and immunodiagnostic reagent set according to the manufacturer's protocol.

SOFA and APACHE II scales were used for comprehensive assessment of clinical status and risk of adverse outcomes. In the course of treatment, adverse reactions during the procedures and final outcome of the hospital stay (duration of stay in ICU and other departments, 28-day mortality) were assessed.

Hemoperfusion through the Eﬀeron LPS adsorber was performed in hospitalized patients with unstable hemodynamic parameters, obvious signs of septic shock according to SEPSIS-3 (2016), during the ﬁrst hours after making the diagnosis of septic shock. The procedures were performed on MultiFiltrate (Fresenius) along the veno-venous bypass. After LPS-selective hemoperfusion procedure, continuous veno-venous hemodiaﬁltration (CVVHDF) was performed on MultiFiltrate (Fresenius).

Statistical analysis. Statistical analysis of research data was carried out using descriptive statistics. The test for normal distribution of paired variable changes before and after hemosorption was performed for each data group using the Shapiro-Wilk test, the hypothesis of normal distribution was rejected at P<0.05. To assess the statistical signiﬁcance of diﬀerences between groups, in distribution diﬀering from the normal, the bilateral Wilcoxon test for paired samples or Mann-Witney test for independent groups were used. In normal distribution of paired variable changes in groups, the signiﬁcance of differences was assessed using the Student's paired bilateral t-criterion. The value of P<0.05 was taken as the cutoﬀ value for statistical signiﬁcance. When comparing groups by categories of treatment outcome "survived-dead" in the group of patients undergoing hemosorption and the group of patients with abdominal sepsis who did not get hemosorbents (control sample), the exact Fisher's test and the calculation of sample power adequacy at alpha=0.05 were used (SigmaPlot 12.5, Systat Software,USA). The Fisher test was also used to compare the percentage of abdominal sepsis and the sex distribution between the above-mentioned groups of patients.

The ultimate goal of the study was to improve treatment outcomes in patients with septic shock and acute renal failure through combined use of LPS-selective hemoperfusion and prolonged venovenous hemodiaﬁltration.

ELIGIBILITY:
Inclusion Criteria:

1. Gram-negative agents in the blood; or detection of an infection focus suggesting Gram-negative agents; or suspected infection based on patient condition, presence of at least two criteria for a systemic inﬂammatory response and procalcitonin (PCT) level ≥ 2 ng/ml;
2. severity of organ dysfunction assessed on a Sepsis-related Organ Failure Assessment (SOFA) scale > 4 points as a result of an evident or suspected infection;
3. need for vasopressor support after administration of ﬂuids to maintain an average blood pressure of at least 65 mmHg. and lactate level in serum > 2 mmol/l (optional, for diagnosis of septic shock).

An additional criterion was the endotoxin activity exceeding 0.6 units according to EAA

Exclusion Criteria:

* terminal condition,
* ongoing internal bleeding or high risk of bleeding,
* severe heart failure (left ventricular ejection fraction < 25%),
* decompensated liver failure,
* body weight less than 20 kg,
* age < 18 or > 80 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included 9 surgical patients with clinical signs of septic shock (SEPSIS-3, 2016) who were admitted to the intensive care unit (ICU) in 2019-2020.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Effect of Efferon LPS hemoperfusion on vasopressor dose after initiation of use in patients with abdominal sepsis complicated by septic shock. | 1-120 hours
  The time (number of hours) from inclusion in the study to the earliest time that the 'resolution of septic shock' event is achieved. Event criteria is end of vasopressor support (persistence of effect - for 4 hours).

SECONDARY OUTCOMES:
Effect of the Efferon LPS hemoperfusion on pulmonary oxygen metabolism function in patients with abdominal sepsis complicated by septic shock | 1-120 hours
  Value of oxygenation index (Pa02 / Fi02 (Pa) every 24 hours ± 1 hour from the start of hemoperfusion (hour 0) to 120 hours.
Effect of LPS Efferon hemoperfusion on SOFA scores in patients with abdominal sepsis complicated by septic shock. | 1-120 hours
  Value of indicators on the SOFA scale every 24 hours ± 1 hour from the start of hemoperfusion (hour 0) to 120 hours.
Effect of LPS Efferon hemoperfusion on procalcitonin levels in patients with abdominal sepsis complicated by septic shock. | 1-120 hours
  Value of procalcitonin levels every 24 hours ± 1 hour from the start of hemoperfusion (hour 0) to 120 hours
Effect of LPS Efferon hemoperfusion on endotoxin activity in patients with abdominal sepsis complicated by septic shock. | 1-72 hours
  Value of endotoxin levels every 24 hours ± 1 hour from the start of hemoperfusion (hour 0) to 72 hours
Effect of LPS Efferon hemoperfusion on IL-1β levels in patients with abdominal sepsis complicated by septic shock. | 1-24 hours
  Value of IL-1β levels from the start of hemoperfusion (hour 0) to 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Timur Kim, MD, Principal Investigator — N.I. Pirogov Clinical City Hospital No. 1
Locations (1):
- N.I. Pirogov City Clinical Hospital No. 1, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Seymour CW, Liu VX, Iwashyna TJ, Brunkhorst FM, Rea TD, Scherag A, Rubenfeld G, Kahn JM, Shankar-Hari M, Singer M, Deutschman CS, Escobar GJ, Angus DC. Assessment of Clinical Criteria for Sepsis: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):762-74. doi: 10.1001/jama.2016.0288. PMID 26903335
- [Result] Besen BAMP, Romano TG, Nassar AP Jr, Taniguchi LU, Azevedo LCP, Mendes PV, Zampieri FG, Park M. Sepsis-3 definitions predict ICU mortality in a low-middle-income country. Ann Intensive Care. 2016 Dec;6(1):107. doi: 10.1186/s13613-016-0204-y. Epub 2016 Nov 2. PMID 27807819
- [Result] Hurley JC. The Role of Endotoxin in Septic Shock. JAMA. 2019 Mar 5;321(9):902-903. doi: 10.1001/jama.2018.20874. No abstract available. PMID 30835303
- [Result] Shoji H, Tani T, Hanasawa K, Kodama M. Extracorporeal endotoxin removal by polymyxin B immobilized fiber cartridge: designing and antiendotoxin efficacy in the clinical application. Ther Apher. 1998 Feb;2(1):3-12. doi: 10.1111/j.1744-9987.1998.tb00066.x. PMID 10227782
- [Result] Zhou F, Peng Z, Murugan R, Kellum JA. Blood purification and mortality in sepsis: a meta-analysis of randomized trials. Crit Care Med. 2013 Sep;41(9):2209-20. doi: 10.1097/CCM.0b013e31828cf412. PMID 23860248
- [Result] Cruz DN, Perazella MA, Bellomo R, de Cal M, Polanco N, Corradi V, Lentini P, Nalesso F, Ueno T, Ranieri VM, Ronco C. Effectiveness of polymyxin B-immobilized fiber column in sepsis: a systematic review. Crit Care. 2007;11(2):R47. doi: 10.1186/cc5780. PMID 17448226
- [Result] Esteban E, Ferrer R, Alsina L, Artigas A. Immunomodulation in sepsis: the role of endotoxin removal by polymyxin B-immobilized cartridge. Mediators Inflamm. 2013;2013:507539. doi: 10.1155/2013/507539. Epub 2013 Oct 22. PMID 24249974
- [Result] Yaroustovsky M, Abramyan M, Krotenko N, Popov D, Plyushch M, Rogalskaya E, Nazarova H. Combined extracorporeal therapy for severe sepsis in patients after cardiac surgery. Blood Purif. 2014;37(1):39-46. doi: 10.1159/000357015. Epub 2014 Feb 5. PMID 24503765
- [Result] Yaroustovsky M, Abramyan M, Popok Z, Nazarova E, Stupchenko O, Popov D, Plushch M, Samsonova N. Preliminary report regarding the use of selective sorbents in complex cardiac surgery patients with extensive sepsis and prolonged intensive care stay. Blood Purif. 2009;28(3):227-33. doi: 10.1159/000231988. Epub 2009 Aug 14. PMID 19684388
- [Result] Martin EL, Cruz DN, Monti G, Casella G, Vesconi S, Ranieri VM, Ronco C, Antonelli M. Endotoxin removal: how far from the evidence? The EUPHAS 2 Project. Contrib Nephrol. 2010;167:119-125. doi: 10.1159/000315926. Epub 2010 Jun 1. PMID 20519906
- [Result] Iba T, Klein DJ. The wind changed direction and the big river still flows: from EUPHRATES to TIGRIS. J Intensive Care. 2019 May 16;7:31. doi: 10.1186/s40560-019-0386-0. eCollection 2019. PMID 31131109
- [Result] Yin C, Liu W, Liu Z, Huang Y, Ci L, Zhao R, Yang X. Identification of potential serum biomarkers in pigs at early stage after Lipopolysaccharide injection. Res Vet Sci. 2017 Apr;111:140-146. doi: 10.1016/j.rvsc.2017.02.016. Epub 2017 Feb 17. PMID 28249176
- [Result] Kogelmann K, Jarczak D, Scheller M, Druner M. Hemoadsorption by CytoSorb in septic patients: a case series. Crit Care. 2017 Mar 27;21(1):74. doi: 10.1186/s13054-017-1662-9. PMID 28343448